CLINICAL TRIAL: NCT03389542
Title: Randomized Comparison of Early Mitral ValvE Repair Versus Watchful Waiting for Asymptomatic SEvere Degenerative Mitral Regurgitation Due to Leaflet Prolapse
Brief Title: Early Mitral ValvE Repair Versus Watchful Waiting for Asymptomatic SEvere Degenerative Mitral Regurgitation
Acronym: REVERSE-MR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2017_843_0005; 2017-A00364-49 (Registry Identifier: ID-RCB number)
Record Dates: First submitted 2017-12-26; First posted 2018-01-03 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Degenerative Mitral Regurgitation (MR) Due to Leaflet Prolapse
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early mitral valve repair (Experimental): Surgery will be performed within 3 months after randomization. Clinical interview will be performed at discharge, at 6 months and afterwards yearly until the end of follow-up. Echocardiography will be performed at discharge, at 6 months and at the end of follow-up.
  Interventions: Procedure: Surgery
- Conservative management (Active Comparator): Patients will be followed up by clinical interview and echocardiography every 6 months.
  Interventions: Other: Clinical interview and echocardiography

INTERVENTIONS:
Procedure: Surgery — Early mitral valve repair
  Arms: Early mitral valve repair
Other: Clinical interview and echocardiography — Clinical interview and echocardiography every 6 months.
  Arms: Conservative management

SUMMARY:
Degenerative mitral regurgitation (MR) due to leaflet prolapse is frequent and can be surgically repaired in the vast majority of patients. Despite the efficacy of mitral valve repair, an ongoing international controversy exists regarding the need to perform early surgery in asymptomatic patients with severe MR and no sign of LV dysfunction in whom the probability of successful and durable repair is very high. In this group of patients, differing views of the risks of uncorrected severe MR exist: considered as benign by those supporting medical "watchful waiting" or associated with significant excess mortality/morbidity by those advocating early surgery. This controversy can only be resolved by a randomized controlled trial which is still lacking.

The main objective is to demonstrate the superiority of early mitral valve repair in patients with asymptomatic severe MR due to leaflet prolapse compared to an initial conservative management in terms of all-cause death and cardiovascular morbidity during five years follow-up.

DETAILED DESCRIPTION:
Experimental group: In patients randomized to early mitral valve repair, surgery will be performed within 3 months after randomization. Clinical interview will be performed at discharge, at 6 months and afterwards yearly until the end of follow-up. Echocardiography will be performed at discharge, at 6 months and at the end of follow-up.

Control group: Patients randomized to initial conservative management will be followed up by clinical interview and echocardiography every 6 months. Patients will be instructed to report any change in functional status in a prompt manner. Surgery will be indicated at the onset of symptoms or if one or more of the following occur during follow-up: LV end-systolic diameter >40mm, LV ejection fraction <60%, recurrent atrial fibrillation, or resting systolic pulmonary artery pressure >50mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic patients according history or an exercise test in those able to perform it if there is a doubt about the absence of symptoms
* Severe (grade IV) degenerative MR due to leaflet prolapse assessed by echocardiography
* LV ejection fraction by Simpson biplane method ≥60% and LV end-systolic diameter by TM echocardiography ≤40mm
* Sinus rhythm on the inclusion ECG
* Pulmonary artery pressure ≤50 mmHg by Doppler echocardiography.
* High probability of mitral valve repair
* EuroSCORE II ≤ 3%

Exclusion Criteria:

* Mitral stenosis or > mild aortic valve disease (stenosis or regurgitation)
* Congenital heart disease (except patent foramen ovale or atrial septal defect)
* Patients with cardiac prostheses
* Previous myocardial infarction
* Previous cardiac surgery
* Extra cardiac comorbidity with life expectancy < 5 years
* Recent history of psychiatric disease (including drug or alcohol abuse)
* Therapy with an investigational intervention at the time of screening or plan to enrol patient in additional intervention study during participation in this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
death and occurrence of adverse cardiovascular events | during 5 years
  Time from randomization to the first occurrence of one of the following composite end-point including all-cause death and occurrence of adverse cardiovascular events (heart failure, atrial fibrillation, infective endocarditis, cerebrovascular events).

CONTACTS AND LOCATIONS:
Overall Officials: Christophe TRIBOUILLOY, MD, PhD, Principal Investigator — CHU Amiens
Locations (2):
- France (2):
  - CHU Amiens-Picardie, Amiens
  - Centre Cardiologique du Nord, Saint-Denis